CLINICAL TRIAL: NCT01906554
Title: Determining Whether or Not Egg Ingestion Increases Concentrations of Trimethylamine N-oxide (TMAO) in Plasma and Urine and Activates LDL Oxidation in Humans
Brief Title: Plasma and Urine TMAO Formation and Changes to Oxidized LDL After Ingestion of Different Amounts of Egg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Steven Zeisel, Professor of Nutrition and Pediatrics, Director, UNC Nutrition Research Institute, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: A12-1066-001
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Biomarkers of Cardiovascular Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- Egg Dose (Experimental)
  Interventions: Other: Egg Dose

INTERVENTIONS:
Other: Egg Dose — Different quantities of eggs

SUMMARY:
Eggs contain an essential nutrient called choline and adequate levels of choline are required for good health. Studies in mice have demonstrated that high levels of choline may increase risk of heart disease through a process that involves the breakdown of choline by gut bacteria. Previous research did not show that human consumption of eggs increases risk of heart disease. This study is designed to investigate whether the number of eggs in the diet affects blood and urine markers for heart disease.

DETAILED DESCRIPTION:
Diets low in choline have adverse health consequences, while observations in humans and experiments in mouse models suggest that a diet containing too much choline or phosphatidylcholine may activate inflammatory pathways and increase cardiovascular disease risk through bacterial conversion of choline to trimethylamine (TMA) and its subsequent oxidation to trimethylamine N-oxide (TMAO) in the liver. What is unclear is whether choline and phosphatidylcholine in eggs is a source of TMAO formation, and if so how many eggs must be eaten before enough TMAO is generated to cause increased oxidized LDL (a biomarker for atherosclerosis mechanisms). We hypothesize that TMAO will only be formed from eggs when very large quantities are ingested and that TMAO formation will vary greatly between individuals for any given dietary exposure. This variability will be determined by 1) the dose at which dietary choline or phosphatidylcholine exceeds the absorptive capacity of the volunteer's small intestine and therefore spills into large intestine where gut bacteria have access to it and 2) the bacterial populations that constitute the volunteer's microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* non-smoker
* Body mass index between 20 to 39 kg/m²

Exclusion Criteria:

* History of chronic system disease/s (e.g., hepatic, renal, cardiovascular, intestinal)
* Diabetes controlled by insulin
* Alcohol or illegal drug misuse/abuse
* Use of antibiotics or choline-containing supplements within three months of study
* Allergies to soy, eggs, wheat or other food
* Use of drugs or medications known to alter liver metabolism, cardiovascular and/or kidney function
* Abnormal physical examination or abnormal clinical laboratory values
* Pregnancy
* Unusual dietary habits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of TMAO | TMAO concentrations in plasma collected prior to and 1, 2, 6, 8, and 24 hours after egg ingestion.

SECONDARY OUTCOMES:
Concentration of TMAO in urine | Concentration of TMAO will be measured in 24 hour urine collections that start the morning of the egg dose

OTHER OUTCOMES:
Changes to plasma oxidized LDL | Oxidized LDL will be measured in plasma collected prior to and 24 hours after ingestion of each egg dose

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Zeisel, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill Nutrition Research Institute, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Miller CA, Corbin KD, da Costa KA, Zhang S, Zhao X, Galanko JA, Blevins T, Bennett BJ, O'Connor A, Zeisel SH. Effect of egg ingestion on trimethylamine-N-oxide production in humans: a randomized, controlled, dose-response study. Am J Clin Nutr. 2014 Sep;100(3):778-86. doi: 10.3945/ajcn.114.087692. Epub 2014 Jun 18. PMID 24944063